CLINICAL TRIAL: NCT06499792
Title: Effectiveness of the Transversus Abdominis Plane Block (TAP-Block) Associated With Opioid Spinal Anesthesia on Analgesia After Cephalic Duodenopancreatectomy
Brief Title: Effectiveness of the Transversus Abdominis Plane Block Associated With Opioid Spinal Anesthesia on Analgesia After Cephalic Duodenopancreatectomy
Acronym: DPC-RATAP
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9134
Record Dates: First submitted 2024-07-05; First posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic Cancer; Cephalic duodenopancreatectomy; Transversus Abdominis Plane Block; TAP Bloc
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Duodenopancreatectomy is a major, risky surgery that causes significant post-operative pain. Optimizing perioperative analgesia remains a challenge, and requires multimodal management, notably involving locoregional analgesic techniques.

The thoracic epidural helps reduce perioperative pain, as well as certain postoperative complications. However, epidural analgesia is not without effects, and the data remains quite heterogeneous depending on the studies regarding its benefits and risks: more frequent hypotension, significant technical failures, length of hospitalization depending on the series, marginal benefit clinically of little relevance... And the existence of contraindications to the epidural such as the performance of vascular resections requiring curative intraoperative anticoagulation also limit its daily use.

The search for alternatives to the epidural in this context has seen the emergence of the use of intrathecal injection of Morphine and the performance of TAP Block perioperatively for duodenopancreatectomies. Morphine spinal anesthesia is an analgesic technique that is simpler and just as effective as the thoracic epidural. The TAP Block has also proven its effectiveness in major colorectal surgeries.

The literature on the subject remains poor and very few studies have focused on alternatives to thoracic epidurals. If the superiority of TAP Block and spinal anesthesia have been evaluated in isolation, no study has yet compared the effectiveness of the combination of TAP Block-Spinal anesthesia compared to that of TAP Block alone in the management of post pain. duodenopancreatectomy.

At the Strasbourg University Hospital, the Anesthesia team in hepatic and pancreatic surgery made a change in practice in June 2023: from a TAP Block, the team performs a TAP-Block combined with a unique Morphinic spinal anesthesia preoperatively for cephalic duodenopancreatectomy (CDP). The objective of the study is to evaluate the effectiveness and safety of this change in practice.

ELIGIBILITY:
Inclusion Criteria:

* Major subject (≥18 years old)
* Planned cephalic or total duodeno-pancreatectomy surgery, associated or not with additional vascular procedures or liver resections by laparotomy, at the Strasbourg University Hospital for the period from June 1, 2022 to May 31, 2024.
* Subject who has not expressed opposition to the reuse of their data for scientific research purposes.

Exclusion Criteria:

* Subject having expressed opposition to participating in the study
* Admission to intensive care following the operation
* Drug addiction withdrawn or not
* Surgery shortened by surgical decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Major subject (≥18 years old) planned cephalic or total duodeno-pancreatectomy surgery, associated or not with additional vascular procedures or liver resections by laparotomy, at the Strasbourg University Hospital for the period from June 1, 2022 to May 31, 2024.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2024-01-03 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Consumption of Morphine in the first 24 hours postoperatively. | Up to 1 year
  Quantitative variables are described using the usual position and dispersion statistics, namely mean, median, minimum, maximum, standard deviation and quantile. The qualitative variables are described with the numbers and proportions of each modality. The Chi2 test will be used to study the crossover between several qualitative variables. The risk of the first kind is set at 5% for all analyses.

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Anesthésiologie - Réanimation Chirurgicale - CHU de Strasbourg - France, Strasbourg, France